CLINICAL TRIAL: NCT03253692
Title: Prospective Multicenter Registry On Radiation Dose Estimates of Cardiac CT Angiography in Daily Practice in 2017 (PROTECTION VI)
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 170146; 17-H-0146
Record Dates: First submitted 2017-08-17; First posted 2017-08-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12-16

CONDITIONS: Coronary Artery Disease; Coronary Disease; Myocardial Ischemia; Arterial Occlusive Diseases; Arteriosclerosis
Keywords: Cardiac Computed Tomography; Radiation; Iterative Reconstruction; Natural History
MeSH Terms: conditions — Coronary Artery Disease; Coronary Disease; Myocardial Ischemia; Arterial Occlusive Diseases; Arteriosclerosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: People ages 18 years and older who need a computed tomography (CT) scan of the heart.

SUMMARY:
Background:

CCTA is a common way to evaluate coronary artery disease. It stands for coronary computed tomography angiography. It uses scanning to look at the arteries that supply blood to the heart. It is noninvasive, widely available, and generally accurate. But it does expose people to radiation. Exposure to high amounts of radiation can increase a person s risk of getting cancer. Researchers want to learn more about the relationship between CCTA and radiation exposure.

Objective:

To see how much radiation is used to take pictures of the heart and how measures to reduce radiation are used around the world.

Eligibility:

People ages 18 years and older who need a computed tomography (CT) scan of the heart

Design:

Participants will be screened with a review of their medical records.

Participants may have a pregnancy test.

Participants will have the scheduled scan. Small, sticky discs will be placed on the chest. A small tube will be placed into a vein in the arm. A contrast material (dye) will be given through it. Participants will lie on the CT scanning table.

A CCTA scan usually takes about 15 minutes if the heart rate is slow and steady.

DETAILED DESCRIPTION:
Cardiac CT angiography is a commonly used test to take detailed pictures of the heart to diagnose heart disease; however, it is associated with radiation exposure. Several technological advances in both scanner hardware and software are now available to reduce the radiation exposure to patients. The purpose of this study is to evaluate the worldwide usage of these radiation dose saving strategies in daily practice and analyze their effect on image quality.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Clinical indication for cardiac CT angiography to evaluate coronary arteries or other cardiac structures
  2. Age equal to or greater than 18 years
  3. Able to understand and willing to sign the Informed Consent Form

EXCLUSION CRITERIA:

1) Female participants who are pregnant or nursing

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Data confirming the inclusion/exclusion criteria will be confirmed at the study visit. Overall, up to 100 subjects will be enrolled locally at the NIH. A member of the study team will review the CT procedures and confirm that the participants do not have any serious health problems or concomitant conditions or medications that would prevent them from having the CT. A member of the study team will perform a pregnancy test (if applicable) in female participants of childbearing potential. If you are nursing, you will be excluded from this study. All tests will follow NIH Clinical Center policies and clinical consent forms for individual tests may be obtained in addition to the study protocol consent as applicable. Sites outside the NIH will use similar standard of care procedures for cardiac CT eligibility.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2017-10-03 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-10-11 (Actual)

PRIMARY OUTCOMES:
Determine radiation dose estimates of cardiac CT angiographies in daily practice | day 0
  We will assess the variation of radiation dose with respect to vendors, CT systems and study sites. Furthermore, we will evaluate the usage of dose saving strategies including the abovementionedin daily practice and analyze their effect on diagnostic image quality. On the basis of the collected data, we will evaluate the potential use of additional dose savings for each individual site.

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Y Chen, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (3):
- United States (3):
  - University of Kentucky, Lexington, Kentucky
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - National Institutes of Health Clinical Center, Bethesda, Maryland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2017-H-0146.html